CLINICAL TRIAL: NCT06509360
Title: How do You Feelee? Does an Ordinary Question a Day Supports Youth in a Forensic Outpatient Setting to Become More Emotional Balanced? A Multiple Case Experimental Design
Brief Title: How do You Feelee? Emotion-based Smartphone App in the Forensic Outpatient Setting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Levvel (Unknown); Arkin (Industry); KFZ-J (Unknown)
Responsible Party: Principal Investigator, Prof. dr. Arne Popma, Prof. dr., Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NL78889.029.22
Record Dates: First submitted 2023-09-01; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Emotion Regulation; Emotional Neglect
Keywords: Smartphone data; Emoji; Emotion regulation; Adolescents; Forensic outpatient care
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Single Case Experimental Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feelee app (Other): Following a Single Case Experimental Design, all participants will follow a ABA baseline: 2-weeks baseline phase without intervention (A), 4-weeks intervention phase using the Feelee app (B) and a 2-weeks follow-up phase without intervention again (B).
  Interventions: Device: Feelee app

INTERVENTIONS:
Device: Feelee app — Adolescents uses the Feelee app for 4-weeks in addition to treatment as usual in the forensic outpatient setting. The use of Feelee involves: submitting one emoji every day and allow the Feelee app to read the following passive data from the health app on the smartphone: number of steps and number of hours of sleep. The collected Feelee data will be presented in a dashboard in the Feelee app itself which will be discussed by the clinician in the weekly treatment session (in case the adolescents agreed to show the Feelee data to the clinician).

SUMMARY:
This intervention study aims to explore the addition of the Feelee app (using active emoji data with passive behavioral data through phone sensing) in treatment as usual for adolescents in the forensic outpatient setting.

Participants will use Feelee for 4 weeks, which means specifying an emoji each day and collecting the passive data on the background. The collected active and passive data will be discussed through the clinicians during the participants' weekly treatment sessions.

DETAILED DESCRIPTION:
Participants will be subjected to a ABA baseline design: including a 2-weeks baseline phase (A), 4-weeks intervention phase (B) and 2-weeks follow-up phase.

During the baseline phase (A), participants will fill in a daily questionnaire that measures different aspects of their emotion regulation skills. The use of the Feelee app is not allowed yet. After 2-weeks, the intervention phase starts, meaning participants will use the Feelee app every day during a 4-weeks period. The use of the Feelee app includes specifying an emoji and collecting the passive data on the background. Furthermore, the collected active and passive data will be discussed through the clinicians during the participants weekly treatment sessions. Participants will also be continuing to complete the daily questionnaire. After 4-weeks, the follow-up phase starts. Participants need to remove the Feelee app and will follow their treatment as usual. However, participants still need to complete the daily questionnaire. After 2-weeks the follow-up phase and main study part has ended.

Throughout the ABA baseline, pre-measurement (T0), post-measurement (T1) follow-up measurement (Tf1) will be conducted before and after the intervention and during follow-up. Last, a 3-months follow-up will be conducted to identify possible long-term effects.

ELIGIBILITY:
Inclusion Criteria:

* At the time of the study in treatment at a forensic outreach youth care organization.
* Expected to be in treatment for at least another 3 months.
* Using a smartphone with Android or IOS operating system.
* Have basic understanding about the use of a smartphone

Exclusion Criteria:

* Adolescents with serious psychiatric problems, such as psychosis or high risk of suicide
* Insufficient understanding of spoken and written Dutch language.
* Adolescents without a smartphone.

Ages: 12 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Emotion regulation: measured by a composite of items from the Difficulties in Emotional Dysregulation Scale (DERS-36) and Regulation of Emotion Systems Survey for daily usage (RESS-EMA) | Daily questionnaire (24 hour interval). From Day 0 (Week 1) up to Day 56 (Week 8).
  Emotion regulation involves the ability to recognize, comprehends and manage emotions.
  The first 2 items are from the DERS-36 scale and measure construct recognize (clarity) and manage (impulse) of emotion regulation. Answers on these scales can be given on a 5-point Likert-scale (0= almost never too 5= almost always).
  The other 4 items are from the RESS-EMA survey The RESS-EMA questionnaire consists of different aspects of the emotion regulation systems and strategies that are suitable for daily usage. The items included in the daily questionnaire are: comprehends (rumination), comprehends (reappraisal), manage (distraction) and manage (suppression). Answers can be given from 0 = not at all to 10 = very much.

SECONDARY OUTCOMES:
Emotional differentiation: Positive and Negative Affect Schedule (PANAS) | Pre-measurement (T0) at Week 1, post-measurement (T1) at Week 6 and follow-up-measurement at Week 8
  Emotional differentiation includes the ability to recognize and distinct different emotional expressions.
  Participants will be asked to rate the extent they experienced one of the 20 items that describes different emotions. The instruments consist of 2 subscales: positive affect and negative affect. These concepts will be scored on a 5-point Likert scale, using the following options: 1 = 'Very slightly/not at all', 2 = 'A little', 3 = 'Moderately', 4 = 'Quite a bit' and 5 = 'Extremely'.
Self-reflection: Self-Reflection and Insight Scale for Youth (SRIS-Y) | Pre-measurement (T0) at Week 1, post-measurement (T1) at Week 6 and follow-up-measurement at Week 8.
  Self-reflection involves the process of looking back at experiences, emotions and behavior in order help individuals to clarify a meaning to it and gain more self-awareness.
  The SRIS-Y is a 17-item self-report questionnaire, answered with a 6-point Likert scale ranging from 1 = 'disagree strongly' to 6= 'agree strongly'. The instrument consists of two subscales self-reflection and and insight resulting in two separate scores. A higher score represents a higher degree of self-reflection and self-insight.
Emotional awareness: Emotional awareness subscale of the Multidimensional Assessment of Interoceptive Awareness (MAIA) | Pre-measurement (T0) at Week 1, post-measurement (T1) at Week 6 and follow-up-measurement at Week 8.
  Emotional awareness involves a subjective understanding of the emotional states and ability to recognize possible causes underlying the emotional states.
  In this study, only the emotional awareness subscale of the MAIA will be used. Answers can be given on a 6-point Likert scale ranging from 0 = 'never' to 5 = 'always'. Scores of the subscale can easily been calculating the total score and dividing it by the number of items belonging to the subscale. A higher score represents a higher degree of emotional awareness.

OTHER OUTCOMES:
Motivation for treatment: Dutch Adolescent Treatment Motivation Questionnaire (ATMQ) | Pre-measurement (T0) at Week 1, post-measurement (T1) at Week 6 and follow-up-measurement at Week 8.
  Motivation for treatment includes the engagement for treatment engagement and willingness to change behavior.
  The ATMQ consists of 11 self-report items with a 3-point Likert scale including 'not true', 'kind of true' and 'true'. The total score is calculated using the average of the number of items. A higher score represents a higher degree of motivation for treatment.
Treatment alliance: Dutch translation of the Working Alliance Inventory (WAV-12) | Pre-measurement (T0) at Week 1, post-measurement (T1) at Week 6 and follow-up-measurement at Week 8.
  Treatment alliance involves the working relationship between client and clinician.
  The WAV-12 questionnaire contains a youth, parental, mentor and family therapist version. In this study only the youth version will be used. The WAV-12 consist of 12 self-report items with a 5-point Likert scale: 1 = 'rarely or never', 2 = 'sometimes', 3 = 'regularly', 4 = 'very often' and 5 = 'always'. Higher scores on this questionnaire indicate a good working alliance between client and clinical.
Evaluation smartphone usage in treatment: the TWente Engagement with E-health Technologies Scales (TWEETS) | Follow-up measurement (Tf1) at Week 8 and 3 months follow-up measurement (Tf2) at Week 21 (3 months after Tf1)
  Evaluation of the smartphone usage in treatment involves the participants experience regarding the usage of the Feelee app in addition to treatment.
  The TWEETS-scale consist of 9 items about engagement of which 3 assess behavioral engagement, 3 cognitive engagement and 3 affective engagement. Answers can be given on a 5-point Likert scale: 0 = 'strongly disagree', 1 = 'disagree', 2 = 'neutral', 3 = 'agree' and 4 = 'strongly agree'
Evaluation usability Feelee app: The System Usability Scale (SUS) | Follow-up measurement (Tf1) at Week 8 and 3 months follow-up measurement (Tf2) at Week 21 (3 months after Tf1)
  Evaluation of the usability of the Feelee app involves the evaluation regarding the user experience (e.g. user interface and design of the app) from participants perspectives.
  The SUS-scale is quick tool to measure usability by 10 items. Answers can be given on a 5-point Likert scale: 0 = 'strongly disagree', 1 = 'disagree', 2 = 'neutral', 3 = 'agree' and 4 = 'strongly agree'.

CONTACTS AND LOCATIONS:
Overall Officials: Arne Popma, Prof. dr., Principal Investigator — Amsterdam UMC, location VUmc
Locations (2):
- Netherlands (2):
  - Inforsa, Amsterdam, North Holland
  - Levvel, Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Dam L, Rietstra S, Van der Drift E, Stams GJJM, Van der Mei R, Mahfoud M, Popma A, Schlossberg E, Pentland A, Reid TG. Can an Emoji a Day Keep the Doctor Away? An Explorative Mixed-Methods Feasibility Study to Develop a Self-Help App for Youth With Mental Health Problems. Front Psychiatry. 2019 Aug 23;10:593. doi: 10.3389/fpsyt.2019.00593. eCollection 2019. PMID 31507464
- [Background] Krasny-Pacini A, Evans J. Single-case experimental designs to assess intervention effectiveness in rehabilitation: A practical guide. Ann Phys Rehabil Med. 2018 May;61(3):164-179. doi: 10.1016/j.rehab.2017.12.002. Epub 2017 Dec 15. PMID 29253607
- [Background] Victor SE, Klonsky ED. Validation of a Brief Version of the Difficulties in Emotion Regulation Scale (DERS-18) in Five Samples. Journal Psychopathologic behavior Assess. 2016; 38(4): 582-589. doi: 10.1007/s10862-016-9547-9
- [Background] Medland H, De France K, Hollenstein T, Mussoff D, Koval P. Regulating emotion systems in everyday life: Reliability and validity of the RESS-EMA scale. European Journal of Psychological Assessment. 2020; 36(3): 437-446. doi:10.1027/1015-5759/a000595
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Sauter FM, Heyne D, Blote AW, van Widenfelt BM, Westenberg PM. Assessing therapy-relevant cognitive capacities in young people: development and psychometric evaluation of the self-reflection and insight scale for youth. Behav Cogn Psychother. 2010 May;38(3):303-17. doi: 10.1017/S1352465810000020. Epub 2010 Apr 12. PMID 20380777
- [Background] Mehling WE, Price C, Daubenmier JJ, Acree M, Bartmess E, Stewart A. The Multidimensional Assessment of Interoceptive Awareness (MAIA). PLoS One. 2012;7(11):e48230. doi: 10.1371/journal.pone.0048230. Epub 2012 Nov 1. PMID 23133619
- [Background] Van der Helm GH, Wissink IB, De Jongh T, Stams GJ. Measuring treatment motivation in secure juvenile facilities. Int J Offender Ther Comp Criminol. 2013 Aug;57(8):996-1008. doi: 10.1177/0306624X12443798. Epub 2012 May 23. PMID 22627687
- [Background] Horvath AO, Greenberg LS. Development and validation of the Working Alliance Inventory. Journal of Counseling Psychology. 1989; 36(2): 223-233. https://doi.org/10.1037/0022-0167.36.2.223
- [Background] Kelders SM, Kip H, Greeff J. Psychometric Evaluation of the TWente Engagement with Ehealth Technologies Scale (TWEETS): Evaluation Study. J Med Internet Res. 2020 Oct 9;22(10):e17757. doi: 10.2196/17757. PMID 33021487
- [Background] Ensink CJ, Keijsers NLW, Groen BE. Translation and validation of the System Usability Scale to a Dutch version: D-SUS. Disabil Rehabil. 2024 Jan;46(2):395-400. doi: 10.1080/09638288.2022.2160837. Epub 2022 Dec 27. PMID 36573399
- [Derived] Leijse MML, van Dam L, Bouwmeester S, van der Pol TM, Breuk R, Popma A. 'I gotta Feeling': Exploring the effects of a smartphone app (Feelee) to enhance adolescents' emotion regulation in forensic outpatient settings: A multiple single-case experimental design. PLoS One. 2026 Feb 6;21(2):e0332111. doi: 10.1371/journal.pone.0332111. eCollection 2026. PMID 41650199
- [Derived] Leijse MML, van Dam L, van der Pol TM, Breuk R, Popma A. The Effects of a Smartphone App (Feelee) to Enhance Adolescents' Emotion Regulation Skills in a Forensic Outpatient Setting: Protocol for a Multiple Single-Case Experimental Design. JMIR Res Protoc. 2025 Jul 2;14:e64756. doi: 10.2196/64756. PMID 40601926
- See also: Website Feelee app — https://www.feelee.nl/en/home
- Available data/document: Individual Participant Data Set — https://www.castoredc.com/ — Individual participant data is collected anonymously in Castor EDC.